CLINICAL TRIAL: NCT00660582
Title: FLOX + Cetuximab (Erbitux®): First Line Treatment for Patients With Metastatic Colorectal Cancer and Wild Type K-RAS Tumor, A Phase II Study
Brief Title: FLOX + Cetuximab (Erbitux®) for Patients With Metastatic Colorectal Cancer and Wild Type K-RAS Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Per Pfeiffer (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Sponsor-Investigator, Per Pfeiffer, Professor, Odense University Hospital
Organization: Odense University Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Nordic 7.5
Record Dates: First submitted 2008-04-11; First posted 2008-04-17 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Erbitux; Colorectal cancer; Oxaliplatin; Flox; Fluorouracil + folinic acid; K-RAS
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cetuximab (Erbitux) — 500 mg/m² every second week, intravenous infusion, 8 cycles
Drug: Oxaliplatin (Eloxatin) + Fluorouracil + folinic acid — Given in combination day 1 and 2, every second week, 8 cycles

SUMMARY:
The Nordic FLOX-regime consists of a combination of bolus 5-FU, leukovorin and oxaliplatin (Eloxatin®). Cetuximab (Erbitux®) is an antibody against the epidermal growth factor receptor (EGFR). The combination of FLOX and weekly Erbitux has been investigated in the Nordic VII study where 571 patients were randomized to FLOX (regime A) or FLOX + Erbitux (regime B or C). Effect-data has not yet been published but the combination is well tolerated, and other studies have shown that Erbitux administered with chemotherapy seem to be more efficient than chemotherapy alone.

The main purpose with this study is to investigate the effect of FLOX and Erbitux given every second week as first line treatment for patients with metastatic colorectal cancer and K-RAS wildtype tumor.

The latest accessible data regarding treatment towards EGFR and K-RAS mutations shows that patients with K-RAS wildtype responds better to treatment than patients with K-RAS mutations.

ELIGIBILITY:
Inclusion Criteria:

Histology and staging disease:

* Histological proven adenocarcinoma of the colon or rectum
* At least one measurable metastatic lesion according to RECIST criteria
* If only one metastatic lesion, histology is mandatory

Mutation level:

* Tumor tissue (primary or metastasis) typological classified as K-RAS wildtype in codon 12 and 13 in exon 1 at real-time PCR

General conditions:

* Age >18 and < 75 years
* WHO performance status ≤ 2; life expectancy of more than 3 months
* Adequate haematological function: (Hb ≥ 6.2 μmol/d, ANC ≥ 1.5 x 109/L, platelets ≥ 100 x 109/L)
* Adequate renal and hepatic functions: total bilirubin ≤ 1.5 upper normal limit, creatinine ≤ 1.25 × upper normal limit, ALAT ≤ 3 x upper normal limits, and ≤ 5 x upper normal limits in case of liver metastases
* Written informed consent prior to randomisation must be obtained and documented according to the local regulatory requirements

Other:

* Fertile patients must use adequate contraceptives

Exclusion Criteria:

Prior therapy:

* Prior chemotherapy for advanced/metastatic disease
* Adjuvant chemotherapy must have ended > 6 months before inclusion
* Prior treatment with Eloxatin
* Prior treatment with Erbitux or other treatment to EGFR

Prior or current history:

* Current indication for resection with a curative intent
* Evidence of CNS metastasis
* Current infection, unresolved bowel obstruction or subobstruction, uncontrolled Crohn's disease or ulcerative colitis
* Current history of chronic diarrhea
* Peripheral neuropathy
* Other serious illness or medical conditions (including contraindication to 5 FU e.g.: angor, myocardial infarction within 6 months, contraindications to monoclonal antibodies)
* Past or concurrent history of malignant neoplasm other than colorectal adenocarcinoma within the past five years, except curatively treated non melanoma skin cancer or in situ carcinoma of the cervix

Concomitant treatments:

* Concomitant (or within 4 weeks before randomisation) administration of any other experimental drug under investigation
* Concurrent treatment with any other anti-cancer therapy

Other:

* Pregnant or breast feeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2008-04; Primary Completion 2011-05 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Per Pfeiffer, MD, Principal Investigator — Odense University Hospital
Locations (6):
- Denmark (3):
  - Department of Oncology, Aalborg University Hospital, Aalborg
  - Department of Oncology, Herlev University Hospital, Herlev
  - Department of Oncology, Odense University Hospital, Odense
- Norway (2):
  - Department of Oncology, Haukeland University Hospital, Bergen
  - Kreftsenteret, Ullevaal University Hospital, Oslo
- Section of Oncology, Uppsala University Hospital, Uppsala, Sweden